CLINICAL TRIAL: NCT01424735
Title: Outcomes of TLR-9 Antagonism in Steroid Resistant Optic Neuritis; A Pilot Study
Brief Title: TLR-9 Antagonism in Steroid Resistant Optic Neuritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sudhalkar Eye Hospital (Other)
Responsible Party: Principal Investigator, Aditya Sudhalkar, Dr. Aditya Sudhalkar, Sudhalkar Eye Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21234EH
Record Dates: First submitted 2011-08-25; First posted 2011-08-29 (Estimated); Last update posted 2011-08-29 (Estimated); Status verified 2011-08

CONDITIONS: Optic Neuritis
Keywords: Best corrected Visual Acuity; Pupillary Reaction; Colour vision; Disc edema
MeSH Terms: conditions — Optic Neuritis; Pupil Disorders | interventions — Immuvac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mw. (Experimental): Administration of immunomodulator Mw.
  Interventions: Drug: Mycobacterium w.(Mw)-freeze dried extract 0.5ml

INTERVENTIONS:
Drug: Mycobacterium w.(Mw)-freeze dried extract 0.5ml — 0.5 ml of Mw in 500ml 0.9% normal saline administered over two hours as an infusion. 2ml(4mg/ml) of dexamethasone administered two hours prior to Mw administration
  Other Names: IMMUVAC

SUMMARY:
Although idiopathic steroid resistant optic neuritis is very uncommon, there is no established treatment protocol for such patients. Toll like receptors (TLRs) especially TLR-9 has been shown to play a role in the pathogenesis of optic neuritis. This small case series aims to determine whether immunomodulators directed specifically at TLR-9(i.e. TLR-9 antagonism)play any role in improving the visual function in such patients.

ELIGIBILITY:
Inclusion Criteria:

Unilateral Steroid Resistant Optic Neuritis

Exclusion Criteria:

* bilateral optic neuritis
* Associated Systemic disease
* Prior treatment received

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2006-07; Primary Completion 2010-01 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Improvement in all aspects of visual function | upto 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bakulesh M Khamar, M.S. Ophthalmology, Principal Investigator — Thakore Eye Hospital, Ahmedabad; Mayuri B Khamar, M.S.Ophthalmology, Principal Investigator — M & J Institute Of Ophthalmology
Locations (1):
- Sudhalkar Eye Hospital, Vadodara, Gujarat, India